CLINICAL TRIAL: NCT01094717
Title: A Comparison of Treatment of Psoriasis With Acitretin or Tazarotene Gel 0.1% and Active or Sham Treatments With the 308 nm Excimer Laser
Brief Title: Acitretin or Tazarotene Gel and Excimer Laser for Treatment of Psoriasis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of efficacy and lack of funding
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kristina Callis, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB_00031865
Record Dates: First submitted 2010-03-25; First posted 2010-03-29 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Psoriasis
Keywords: psoriasis; excimer; acitretin; tazarotene
MeSH Terms: conditions — Psoriasis | interventions — Acitretin; Lasers, Excimer; tazarotene

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Excimer laser active and comparator were delivered the same way by a non-blinded person who applies a cap to the laser head to block UV rays for a sham administration. The masking was done by blindfolding the patients so they could not see which side was treated with active or sham laser. The outcomes assessor did their assessment in a separate room and access restricted to the randomization assignments.
Oversight: Data Monitoring Committee: No

ARMS (4):
- acitretin and active excimer laser (Experimental): patients enrolled in the acitretin arm will be treated with acitretin 25 mg daily and excimer (active) to randomly assigned left or right side of body psoriasis lesions.
  Interventions: Drug: Acitretin 25Mg Oral Capsule; Device: Excimer laser
- acitretin and sham excimer laser (Experimental): Patients in this arm were treated with acitretin 25 mg daily and sham (placebo) excimer laser to randomly assigned left or right side of body psoriasis lesions.
  Interventions: Drug: Acitretin 25Mg Oral Capsule; Device: Sham excimer laser
- tazarotene and active excimer laser (Experimental): patients enrolled in this arm were treated with tazarotene 0.1% gel topical application daily and excimer (active) laser to randomly assigned left or right side of body psoriasis lesions.
  Interventions: Device: Excimer laser; Drug: Tazarotene 0.1% Gel,Top
- tazarotene and sham excimer laser (Experimental): patients enrolled in this arm were treated with tazarotene 0.1% gel topical application daily and sham excimer laser to randomly assigned left or right side of body psoriasis lesions.
  Interventions: Drug: Tazarotene 0.1% Gel,Top; Device: Sham excimer laser

INTERVENTIONS:
Drug: Acitretin 25Mg Oral Capsule — Acitretin 25 mg oral daily for 12 weeks
  Arms: acitretin and active excimer laser; acitretin and sham excimer laser
Device: Excimer laser — Lesions on randomly assigned left or right side of body were treated with 308nm excimer laser.
  Arms: acitretin and active excimer laser; tazarotene and active excimer laser
Drug: Tazarotene 0.1% Gel,Top — Topical tazarotene 0.1% gel was applied daily to active lesions.
  Arms: tazarotene and active excimer laser; tazarotene and sham excimer laser
Device: Sham excimer laser — Lesions on randomly assigned left or right side of body were treated with sham excimer laser (opaque cover on the laser device).
  Arms: acitretin and sham excimer laser; tazarotene and sham excimer laser

SUMMARY:
This is a randomized, double-blind study of excimer (308-nm UVB) laser added to either tazarotene 0.1% gel or acitretin 25 mg daily for plaque psoriasis.

The primary objective of this study is to compare the improvement of psoriatic plaques with and without excimer laser (308-nm UVB) treatment, applied in a randomized and blinded fashion, in subjects on acitretin 25 mg or tazarotene gel 0.1% QD.

DETAILED DESCRIPTION:
The hypothesis of this study is that excimer (308-nm UVB) laser added to either tazarotene 0.1% gel or acitretin 25 mg daily will lead to improved efficacy of these treatments alone.

The primary objective of this study is to compare the improvement of psoriatic plaques with and without excimer laser (308-nm UVB) treatment, applied in a randomized and blinded fashion, in subjects on acitretin 25 mg or tazarotene gel 0.1% QD. The primary endpoint will be the comparison between the change in NPF score of plaques treated with excimer laser and those treated with sham treatment.

The secondary objectives are to compare the number of excimer light treatments and time necessary to achieve an average lesion assessment score of 0 to 1 in subjects treated with acitretin 25 mg PO or tazarotene gel 0.1% QD, and to evaluate adverse events related to combinations of the study treatments.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent
* Must be at least 18 years old
* Must have been diagnosed with stable plaque type psoriasis covering between 1 and 5% BSA
* NPF-PS ≥8 (based additive scores averaged over all lesions for erythema, scale, and thickness range of score = 0-5)
* No systemic or phototherapy in the 4 wks prior to entering the study
* No topical therapy other than emollients (no corticosteroids, vitamin D analogs, vitamin A analogs) in the 2 wks prior to entering the study
* Women on tazarotene gel must not be pregnant nor planning to become pregnant during the study and must be on two forms of birth control
* Subjects known to not tolerate oral acitretin at 25 mg/day and women of child-bearing potential may be enrolled and treated with topical tazarotene gel 0.1%

Exclusion Criteria:

Candidates will be excluded from study entry if any of the following exclusion criteria exist at the time of enrollment:

* Unstable disease
* Only treatable sites are in intertriginous areas or on face
* Subjects unable to tolerate frequency of visits
* NPF-PS severity score <8 additive score of erythema, scale, and thickness, averaged over all lesions
* History of inability to tolerate topical tazarotene 0.1% gel and or acitretin 25 mg/day
* Women of childbearing potential are excluded from the actretin arm of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristina C Duffin, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Department of Dermatology, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acitretin and Excimer: Patients treated with acitretin 25 mg daily and active excimer laser to lesions on one half of the body (side assigned to active laser) and sham excimer laser (opaque cover on laser lens)to lesions on the other half of the body (side assigned to sham laser).
- Tazarotene Gel and Excimer Laser: patients in this group applied tazarotene 0.1% gel to all lesions and active excimer laser used to treat lesions on one half of the body (side assigned to active laser) and sham excimer laser (opaque cover applied over laser lens) used to treat lesions on the other half of the body (side assigned to sham laser).
Period: Overall Study
Arm/Group | Acitretin and Excimer | Tazarotene Gel and Excimer Laser
Started | 3 | 10
Completed | 3 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acitretin and Excimer; Tazarotene and Excimer: excimer vs sham excimer: half of lesions will be treated with excimer laser; half of lesions will be treated with sham excimer (opaque cover on the laser device)
- Total: Total of all reporting groups
Arm/Group | Acitretin and Excimer | Tazarotene and Excimer | Total
Number analyzed (Participants) | 3 | 10 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 8 | 10
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (19.4) | 46.4 (17.2) | 46.6 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 4
  Male | 3 | 6 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 10 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in the NPF Psoriasis Score of Plaques
Description: mean % change in the National Psoriasis Foundation (NPF) psoriasis score of the target plaques [higher percent change in NPF score is consistent with improvement, while higher absolute NPF score is consistent with worse disease, minimum score of 0 (no disease) and maximum score of 30 (worst disease)]
Time Frame: week 8
Measure: Mean (Standard Deviation); unit: percentage change
Groups:
- Acitretin and Excimer: patients received acitretin 25 mg daily and active excimer laser excimer twice weekly to lesions on one of half of the body that was assigned to active laser (left or right determined by randomization)
- Acitretin and Sham (Placebo) Excimer: patients received acitretin 25 mg daily and sham (placebo) excimer twice weekly to lesions on one of half of the body that was assigned to sham (left or right determined by randomization)
- Tazarotene Gel and Excimer Laser: patients received topical tazarotene gel 0.1% applied to all lesions daily, and active excimer laser excimer twice weekly to lesions on one of half of the body that was assigned to active laser (left or right determined by randomization)
- Tazarotene Gel and Sham (Placebo) Excimer: patients receive tazarotene gel 0.1% applied daily to all lesions, and sham excimer twice weekly to lesions on one of half of the body that was assigned to sham (left or right determined by randomization)
Arm/Group | Acitretin and Excimer | Acitretin and Sham (Placebo) Excimer | Tazarotene Gel and Excimer Laser | Tazarotene Gel and Sham (Placebo) Excimer
Number analyzed (Participants) | 3 | 3 | 10 | 10
percentage change | -64.0 (26.5) | -52.1 (36.3) | -32.7 (10.4) | -26.9 (12.8)

2. Secondary Outcome: Number of Patients That Achieved an Average Lesion Assessment Score of 0 or 1 at Week 12.
Description: number of patients who achieved average lesion assessment score of 0 or 1 by the Target Plaque Sum Score (TPSS) for each arm/intervention. For the TPSS, the target plaque was assessed separately for induration, scaling, and erythema using a 6-point severity scale (0 = none and 5 = severe) and the scores were summed to produce the Target Plaque Sum Score [15-point scale; maximum (most severe) score 15].
Time Frame: 8 weeks
Measure: Number; unit: participants
Groups:
- Acitretin and Excimer: patients enrolled in the acitretin arm will be treated with acitretin 25 mg daily and excimer (active) to one side of the body and sham excimer (placebo) to the to the other side of body.
  excimer vs sham excimer: half of lesions will be treated with excimer laser; half of lesions will be treated with sham excimer (opaque cover on the laser device)
- Acitretin and Sham Excimer Laser: patients treated with acitretin 25 mg and sham excimer laser.
- Tazarotene and Excimer: patients enrolled in the tazarotene arm will be treated with topical tazarotene 0.1% gel and excimer (active) to one side of the body and sham excimer (placebo) to the to the other side of body.
  excimer vs sham excimer: half of lesions will be treated with excimer laser; half of lesions will be treated with sham excimer (opaque cover on the laser device)
- Tazarotene and Sham Excimer Laser: patients receiving tazotene gel 0.1% and sham excimer laser to half of body.
Arm/Group | Acitretin and Excimer | Acitretin and Sham Excimer Laser | Tazarotene and Excimer | Tazarotene and Sham Excimer Laser
Number analyzed (Participants) | 3 | 3 | 10 | 10
participants | 1 | 0 | 0 | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: We will collect number and types of adverse events for the excimer-treated vs. sham-treated sites
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Acitretin and Active Excimer Laser: patients enrolled in the acitretin arm will be treated with acitretin 25 mg daily and excimer (active) to randomly assigned left or right side of body psoriasis lesions.
  excimer laser (active): Lesions on randomly assigned left or right side of body were treated with active excimer laser by an increasing dose level per a standard of care protocol.
  Acitretin 25 MG: Patients assigned to this intervention took oral acitretin 25 mg daily.
- Acitretin and Sham Excimer Laser: Patients in this arm were treated with acitretin 25 mg daily and sham (placebo) excimer laser to randomly assigned left or right side of body psoriasis lesions.
  excimer laser (sham): Lesions on randomly assigned left or right side of body were treated with sham excimer laser (opaque cover on the laser device).
  Acitretin 25 MG: Patients assigned to this intervention took oral acitretin 25 mg daily.
- Tazarotene and Active Excimer Laser: patients enrolled in this arm were treated with tazarotene 0.1% gel topical application daily and excimer (active) laser to randomly assigned left or right side of body psoriasis lesions.
  excimer laser (active): Lesions on randomly assigned left or right side of body were treated with active excimer laser by an increasing dose level per a standard of care protocol.
  Tazarotene 0.1% gel: Patients assigned to this intervention applied topical tazarotene gel 0.1% to all lesions daily.
- Tazarotene and Sham Excimer Laser: patients enrolled in this arm were treated with tazarotene 0.1% gel topical application daily and sham excimer laser to randomly assigned left or right side of body psoriasis lesions.
  excimer laser (sham): Lesions on randomly assigned left or right side of body were treated with sham excimer laser (opaque cover on the laser device).
  Acitretin 25 MG: Patients assigned to this intervention took oral acitretin 25 mg daily.
Arm/Group | Acitretin and Active Excimer Laser | Acitretin and Sham Excimer Laser | Tazarotene and Active Excimer Laser | Tazarotene and Sham Excimer Laser
Number analyzed (Participants) | 3 | 3 | 10 | 10
Participants
  any adverse event | 2 | 2 | 4 | 4
  severe adverse events | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Acitretin and Excimer | Tazarotene and Excimer
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 2/3 | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acitretin and Excimer (N=3) | Tazarotene and Excimer (N=10)
Dry lips (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Dry eyes (Eye disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Rigors (General disorders) | 1 (1) | 0 (0)
Bump on figner (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Elevated triglycerides (Endocrine disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3)
Inflamed seborrheic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes